CLINICAL TRIAL: NCT02928003
Title: Chronic Neuropathic Pain After Lung Surgery: Prevalence and Predictive Factors
Acronym: DOLORPOUMON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015/35; 2016-A00045-46 (Other: ANSM)
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Pain
Keywords: Lung surgery
MeSH Terms: conditions — Pain | interventions — Pulmonary Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Surgery (Experimental)
  Interventions: Procedure: Lung surgery

INTERVENTIONS:
Procedure: Lung surgery — Genetic analysis and questionnaires

SUMMARY:
Chronic post-thoracotomy pain is the most common long-term complication that occurs after a thoracotomy with a reported incidence of up to 80%. Surgical approach as well as other factors (genetic, psychological) could have a major and independent role in the development of the post operative pain.The main objective of this study is to identify genetic and psychological profile (cognitive and emotional) of patients who develop chronic pain after lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing lung resection surgery.
* 18 years and older (without superior limit);
* Affiliated to french "securité sociale"

Exclusion Criteria:

* Emergency procedure
* litigation or search for compensation;
* Previous intervention in the same region;
* Peripheral neurological pathology (polyneuropathy) or central (brain damage, multiple sclerosis …) that may interfere with the evaluation of the post-operative pain
* Participation in another biomedical research protocol if there is an incompatibility with the present protocol.
* mental disability
* vulnerable person within the meaning of French law,
* poor understanding of French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with chronic pain 4 months after surgery | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Michel-Cherqui, MD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Institut Mutualiste Montsouris, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No